CLINICAL TRIAL: NCT01782313
Title: A Phase II Study of Tivozanib in Patients With Metastatic and Non-resectable Soft Tissue Sarcomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: AVEO Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Mark Agulnik, Principal Investigator, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 12S02; NCI-2012-03188 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STU00073826 (Other: Northwestern University IRB#)
Record Dates: First submitted 2013-01-30; First posted 2013-02-01 (Estimated); Results first posted 2018-08-21 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-08

CONDITIONS: Recurrent Adult Soft Tissue Sarcoma; Stage III Adult Soft Tissue Sarcoma; Stage IV Adult Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — tivozanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (tivozanib) (Experimental): Patients receive tivozanib PO daily on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: tivozanib; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: tivozanib — Given PO
  Other Names: AV-951; oral VEGF receptor tyrosine kinase inhibitor AV-951
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This study is for patients who have been diagnosed with soft tissue sarcoma that has spread (metastasized) or that is not eligible for removal by surgery. The purpose of this study is to determine how soft tissue sarcomas respond to treatment with an investigational drug called tivozanib. In some lab and clinical studies, tivozanib has been shown to interfere with the growth of some types of tumors. The study will also evaluate how safe the study treatment is by observing how many and what kind of adverse events (side effects) participants experience.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the progression-free survival (defined as complete response [CR] + partial response [PR] + stable disease [SD]) assessed at 16 weeks for patients treated with tivozanib.

SECONDARY OBJECTIVES:

I. Overall response rate (defined as CR + PR). II. Clinical benefit rate (CR + PR + SD). III. Overall survival (up to 2 years beyond progression). IV. Correlation of clinical outcome with antibodies for vascular endothelial growth factor receptor 1 (VEGFR1) and VEGFR2.

V. Assess Safety and tolerability.

OUTLINE:

Patients receive tivozanib orally (PO) daily on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity, or until discontinuation per patient preference or physician recommendation.

After completion of study treatment, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed sarcoma of soft tissue
* Patients must have metastatic and/or locally advanced or locally recurrent disease
* Patients must have measurable disease within 4 weeks prior to registration by RECIST 1.1, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral computed tomography (CT) scan; tumor lesions that are situated in a previously irradiated area may be considered measurable for the purposes of this study only if there is evidence of growth of the area following a course of irradiation that cannot be attributed to necrosis or bleeding into the tumor
* Patients must have had a minimum of 1 and a maximum of 4 prior chemotherapy regimens for recurrent/metastatic disease (it will be up to the treating investigator to define what constitutes a "regimen" in each case); the last dose of systemic therapy (include tyrosine kinase inhibitors) must have been given at least 4 weeks prior to initiation of therapy; patients receiving BCNU or mitomycin C must have received their last dose of such therapy at least 6 weeks prior to initiation of therapy
* Patients with brain metastasis that have been treated with definitive surgery or radiation and have been clinically stable for 3 months following the procedure with no neurological signs or symptoms and no requirement for systemic glucocorticoids are eligible for study
* Patients must exhibit an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Absolute neutrophil count >= 1.5 x 10^9/l
* Platelets >= 75 x 10^9/l
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (except for patients with known Gilbert Syndrome)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional ULN
* Serum creatinine =< 1.5 x ULN
* If urine protein:creatinine (UPC) >= 1, then a 24-hour urine protein must be assessed; patients must have a 24-hour urine protein value < 1g to be eligible
* Patients must not have current evidence of another malignancy; there are no restrictions regarding prior history of malignancy
* If female and of childbearing potential, documentation of negative pregnancy test is required within 7 days prior to first dose; sexually active males and females of childbearing potential must agree to use adequate contraceptive measures, while on study and for 30 days after the last dose of study drug; all subjects (and their partners) must agree to use a highly effective method of contraception; effective birth control includes (a) intrauterine device (IUD) plus one barrier method; or (b) 2 barrier methods; effective barrier methods are male or female condoms, diaphragms, and spermicides (creams or gels that contain a chemical to kill sperm)

  * Note: oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions, and are not considered effective for this study
* Adverse events related to prior tumor-specific therapy must have resolved to less than or equal to National Cancer Institute (NCI) Common Terminology Criteria of Adverse Events (CTCAE) (version 4) grade 1 prior to study entry (except alopecia)
* Patients taking cytochrome P450 (CYP)3A4 inducers at the time of screening/registration are still eligible for participation, but whenever possible these medications should be discontinued or changed to one that is not an inducer

  * NOTE: No washout period is required
  * NOTE: It will be up to the treating investigator's discretion to assess whether or not the risk of discontinuing or changing the medication is higher or lower than the risk of continuing it while on study for the individual patient
* Patients must have the ability to understand and the willingness to sign a written informed consent document; signed and dated informed consent must be obtained prior to registration on trial

Exclusion Criteria:

* Patients with any one of the following sarcoma histological subtypes will not be eligible for participation: alveolar soft-part sarcoma, chondrosarcoma, dermatofibrosarcoma, Ewing sarcoma, gastrointestinal stromal tumor (GIST), Kaposi sarcoma, mixed mesodermal tumor/carcinosarcoma, osteosarcoma, and low grade (grade 1) sarcomas; NOTE: Myxoid liposarcoma with t(12;16) or t(22;22) is permitted; rhabdomyosarcoma (Embryonal, Alveolar, pleomorphic), interdigitating dendritic sarcoma, giant cell tumor of bone
* Patients who have had major surgery within 21 days or those who have not recovered from adverse events associated with surgery to =< grade 1 will not be eligible for participation; excluded from such considerations are surgical changes not expected to improve, e.g. removal of muscle tissue; patients may be on replacement glucocorticoids for pre-existing glucocorticoid deficiency (e.g. Addison's disease)
* Patients receiving any other investigational agents will not be eligible for participation
* Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to tivozanib will not be eligible for participation
* Patients with serious and/or unstable pre-existing medical, psychiatric, or other conditions that could interfere with safety, provision of informed consent, or compliance to study procedures and requirements will not be eligible for participation, including but not limited to:

  * Uncontrolled intercurrent illness
  * Ongoing or active infection including HIV, active hepatitis B or C)
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situations that would limit compliance with study requirements will not be eligible for participation
* Pregnant women and women who are breast-feeding will not be eligible for participation
* Patients with a history or clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis will not be eligible for participation; NOTE: Individuals who have previously-treated CNS metastases, are asymptomatic, and have had no requirement for steroids or anti-seizure medications for 3 months prior to first dose of study drug are the exception; screening with CNS imaging studies such as CT or magnetic resonance imaging (MRI) is required only if clinically indicated or if the subject has a history of CNS metastases
* Patients with clinically significant gastrointestinal (GI) abnormalities that may increase the risk for GI bleeding will not be eligible for participation; these include, but are not limited to:

  * Active peptic ulcer disease
  * Known intraluminal metastatic lesion/s with risk of bleeding
  * Inflammatory bowel disease (e.g. ulcerative colitis, Crohn's disease), or other GI conditions with increased risk of perforation
  * History of abdominal fistula, GI perforation, or intra-abdominal abscess within 28 days prior to beginning study treatment
  * Clinically significant (> 1/2 teaspoon) hemoptysis or gastrointestinal hemorrhage in the past 6 months
* Patients with evidence of active bleeding or bleeding diathesis will not be eligible for participation; recent hemoptysis would be >= 1/2 teaspoon of red blood within 8 weeks before first dose of study drug
* Patients with clinically significant GI abnormalities that may affect absorption of investigational product will not be eligible for participation; these include but are not limited to:

  * Malabsorption syndrome
  * Major resection of the stomach or small bowel
* Patients with a corrected QT interval (QTc) > 480 msecs using Bazett's formula (QT Interval / square root(RR interval)) will not be eligible for participation
* Patients with left ventricular ejection fraction (LVEF) < 50% will not be eligible for participation

  * NOTE: patients who do not meet the cutoff for LVEF may be re-screened at a later date and, if eligible then, may be enrolled in the study
* Patients with a history of any one or more of the following cardiovascular conditions within the past 6 months will not be eligible for participation:

  * Cardiac angioplasty or stenting
  * Myocardial infarction
  * Unstable angina
  * Coronary artery bypass graft surgery
  * Symptomatic peripheral vascular disease\
  * Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA)
* Patients with poorly controlled hypertension [defined as systolic blood pressure (SBP) of >= 140 mmHg or diastolic blood pressure (DBP) of >= 90mmHg] will not be eligible for participation

  * Note: Initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry; following antihypertensive medication initiation or adjustment, blood pressure (BP) must be re-assessed three times at approximately 2-minute intervals; at least 24 hours must have elapsed between anti-hypertensive medication initiation or adjustment and BP measurement; these three values will be averaged to obtain the mean diastolic blood pressure and the mean systolic blood pressure; the mean SBP / DBP ratio must be < 140/90 mmHg in order for a subject to be eligible for the study
* Patients with cerebrovascular accident including transient ischemic attack (TIA), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months will not be eligible for participation

  * Note: subjects with recent DVT who have been therapeutically coagulated for at least 6 weeks are eligible
* Patients who had major surgery or trauma within 28 days prior to first dose of investigational product and/or presence of any non-healing wound, fracture, or ulcer (procedures such as catheter placement not considered to be major surgery) will not be eligible for participation
* Patients with known endobronchial lesions and/or lesions infiltrating major pulmonary vessels will not be eligible for participation

  * Note: tumor abutting the vessel is acceptable, but contiguous tumor and vessel is not; CT with contrast is strongly recommended to evaluate such lesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2013-03-06 (Actual); Primary Completion 2015-05-27 (Actual); Study Completion 2016-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Agulnik, MD, Principal Investigator — Northwestern University
Locations (5):
- United States (5):
  - Northwestern University, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- [Derived] Agulnik M, Costa RLB, Milhem M, Rademaker AW, Prunder BC, Daniels D, Rhodes BT, Humphreys C, Abbinanti S, Nye L, Cehic R, Polish A, Vintilescu C, McFarland T, Skubitz K, Robinson S, Okuno S, Van Tine BA. A phase II study of tivozanib in patients with metastatic and nonresectable soft-tissue sarcomas. Ann Oncol. 2017 Jan 1;28(1):121-127. doi: 10.1093/annonc/mdw444. PMID 27771610

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened for accrual on February 25, 2013 with an accrual goal of up to 58 patients. The study was designed to enroll 19 patients initially and and continue to enroll up to 58 patients if 5 or more of the first 19 are progression free at 4 months. The study was closed permanently on February 4, 2015 with 58 patients enrolled.
Period: Reached First Response/Completed 2 Cycle
Arm/Group | Treatment (Tivozanib)
Started | 58
Completed | 52
Not Completed | 6
Not completed — Adverse Event | 3
Not completed — Progressive Disease | 3
Period: Treated Cycle 3
Arm/Group | Treatment (Tivozanib)
Started | 52
Completed | 31
Not Completed | 21
Not completed — Progressive Disease | 21
Period: Treated Cycle 4/Reached 16 Week Response
Arm/Group | Treatment (Tivozanib)
Started | 31
Completed | 25
Not Completed | 6
Not completed — Progressive Disease | 5
Not completed — Adverse Event | 1
Period: Continued Treatment After 16 Weeks
Arm/Group | Treatment (Tivozanib)
Started | 25
Completed | 18
Not Completed | 7
Not completed — Progressive Disease | 6
Not completed — Withdrawal by Subject | 1
Period: Survival Follow up
Arm/Group | Treatment (Tivozanib)
Started | 58
Completed | 57
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Tivozanib)
Number analyzed (Participants) | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 56
  More than one race | 0
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 57
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 58
Prior anti-overexpress vascular endothelial growth factor (VEGF) therapy or anti-VEGF therapy naive [Count of Participants; unit: Participants]
  Prior anti-VEGF therapy | 24
  No prior anti-VEGF therapy | 34

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Progression-free Survival at 16 Weeks.
Description: Progression-free survival from study disease will be evaluated using Response Evaluation Criteria in Solid Tumors (RECIST) Committee, version 1.1 assessed using imaging scans (CT or MRI) and clinical assessment following 16 weeks of treatment.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions", or similar definition as accurate and appropriate.
Time Frame: At 16 weeks of treatment.
Population: 3 patients were not evaluable due to withdrawal tivozanib within the first 14 days of treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Treatment (Tivozanib)
Number analyzed (Participants) | 55
Percentage of patients | 36.4 [23.7 to 49.1]

2. Secondary Outcome: Overall Response Rate Defined as Complete Response and Partial Response.
Description: The response to study treatment will be assessed after every 8 weeks (2 cycles) of therapy using CT or MRI scan images.Overall response rate will be measured per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT or MRI:
  Complete response (CR) = disappearance of all target lesions. Partial Response (PR), = at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD.
Time Frame: Every 2 cycles (8 weeks) up to 2 years
Population: 3 patients were not evaluable due to withdrawal tivozanib within the first 14 days of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Tivozanib)
Number analyzed (Participants) | 55
Participants | 2

3. Secondary Outcome: Clinical Benefit Rate as Defined by Complete Response, Partial Response and Stable Disease.
Description: The clinical benefit of study treatment will be assessed after 8 weeks (2 cycles) of therapy using scanning images (CT or MRI). Clinical benefit rate will be measured per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT or MRI:
  Complete Response (CR) = disappearance of all target lesions. Partial Response (PR), = at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD.
  Progressive Disease (PD) = At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
  Stable Disease (SD) = Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: Every 2 cycles (8 weeks) up to 2 years
Population: 3 patients were not evaluable due to withdrawal tivozanib within the first 14 days of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Tivozanib)
Number analyzed (Participants) | 55
Participants | 32

4. Secondary Outcome: Overall Survival up to 2 Years Beyond Progression
Description: Patients will be followed-up with from first dose of study drug up to 2 years following the date of disease progression.
Time Frame: Time from the first dose of study treatment up to 2 years beyond disease progression
Population: 3 patients were not evaluable due to withdrawal tivozanib within the first 14 days of treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Tivozanib)
Number analyzed (Participants) | 55
Months | 12.2 [8.1 to 16.8]

5. Secondary Outcome: Number of Patients With 0-3 VEGFR1 and VEGFR2 Protein Expression and Time in Days on Treatment
Description: Tissue from biopsy will be collected during screening and proteins (VEGFR1 and VEGFR2) will be evaluated to see if there is a correlation with patient response to treatment.
  VERGFR = vascular endothelial growth factor receptor
  To determine if there was a correlation between response to Tivozanib and VEGFR expression, immunohistochemical (IHC) analysis on archival tumor tissue was performed. We performed standard IHC and applied combined intensity score (from 0 to 3) for antigen expression and proportional score of 0-3 for the cells that were positive. For antigen expression, 0 was no staining, +1 being 1-25% staining, +2 being 26-50% staining and +3 being 50% or greater staining. Number of patients with VEGFR1 expression was correlated with time patients were on treatment in days.
Time Frame: Tissue collected during screening process, prior to first treatment and response measured until 350 days.
Population: 3 patients were not evaluable due to withdrawal tivozanib within the first 14 days of treatment. Not all patients treated on study provided tissue or had sufficient tissue to be analyzed for VEGFR expression.
Measure: Number; unit: participants
Arm/Group | Treatment (Tivozanib)
Number analyzed (Participants) | 40
participants
  VEGFR1 Group 0 : 0 days | 8
  VEGFR1 Group 0 : 50 days | 6
  VEGFR1 Group 0 : 100 days | 2
  VEGFR1 Group 0 : 150 days | 1
  VEGFR1 Group 0 : 200 days | 1
  VEGFR1 Group 0 : 250 days | 1
  VEGFR1 Group 0 : 300 days | 1
  VEGFR1 Group 0 : 350 days | 0
  VEGFR1 Group +1 : 0 days | 3
  VEGFR1 Group +1 : 50 days | 1
  VEGFR1 Group +1 : 100 days | 0
  VEGFR1 Group +1 : 150 days | 0
  VEGFR1 Group +1 : 200 days | 0
  VEGFR1 Group +1 : 250 days | 0
  VEGFR1 Group +1 : 300 days | 0
  VEGFR1 Group +1 : 350 days | 0
  VEGFR1 Group +2 : 0 days | 8
  VEGFR1 Group +2 : 50 days | 4
  VEGFR1 Group +2 : 100 days | 4
  VEGFR1 Group +2 : 150 days | 2
  VEGFR1 Group +2 : 200 days | 0
  VEGFR1 Group +2 : 250 days | 0
  VEGFR1 Group +2 : 300 days | 0
  VEGFR1 Group +2 : 350 days | 0
  VEGFR1 Group +3 : 0 days | 21
  VEGFR1 Group +3 : 50 days | 11
  VEGFR1 Group +3 : 100 days | 4
  VEGFR1 Group +3 : 150 days | 2
  VEGFR1 Group +3 : 200 days | 1
  VEGFR1 Group +3 : 250 days | 1
  VEGFR1 Group +3 : 300 days | 1
  VEGFR1 Group +3 : 350 days | 0
  VEGFR2 Group 0 : 0 days | 19
  VEGFR2 Group 0 : 50 days | 11
  VEGFR2 Group 0 : 100 days | 6
  VEGFR2 Group 0 : 150 days | 2
  VEGFR2 Group 0 : 200 days | 1
  VEGFR2 Group 0 : 250 days | 1
  VEGFR2 Group 0 : 300 days | 1
  VEGFR2 Group 0 : 350 days | 0
  VEGFR2 Group +1 : 0 days | 6
  VEGFR2 Group +1 : 50 days | 4
  VEGFR2 Group +1 : 100 days | 2
  VEGFR2 Group +1 : 150 days | 2
  VEGFR2 Group +1 : 200 days | 1
  VEGFR2 Group +1 : 250 days | 1
  VEGFR2 Group +1 : 300 days | 1
  VEGFR2 Group +1 : 350 days | 0
  VEGFR2 Group +2 : 0 days | 4
  VEGFR2 Group +2 : 50 days | 3
  VEGFR2 Group +2 : 100 days | 0
  VEGFR2 Group +2 : 150 days | 0
  VEGFR2 Group +2 : 200 days | 0
  VEGFR2 Group +2 : 250 days | 0
  VEGFR2 Group +2 : 300 days | 0
  VEGFR2 Group +2 : 350 days | 0
  VEGFR2 Group +3 : 0 days | 8
  VEGFR2 Group +3 : 50 days | 2
  VEGFR2 Group +3 : 100 days | 1
  VEGFR2 Group +3 : 150 days | 0
  VEGFR2 Group +3 : 200 days | 0
  VEGFR2 Group +3 : 250 days | 0
  VEGFR2 Group +3 : 300 days | 0
  VEGFR2 Group +3 : 350 days | 0

6. Secondary Outcome: Treatment Toxicity as Measured by Adverse Events Experienced While on Treatment During Systematic Assessment.
Description: Toxicity will be assessed after 4 weeks (1 cycle) and every 4 weeks during treatment according to the National Cancer Institute's Common Toxicity Criteria for adverse events version 4.0 (CTCAE v4.0). In general adverse events (AEs) will be graded according to the following:
  Grade 1 Mild AE Grade 2 Moderate AE Grade 3 Severe AE Grade 4 Life-threatening or disabling AE Grade 5 Death related to AE
Time Frame: After every 4 weeks (1 cycle) until treatment discontinuation and up to a maximum of 2 years and 10 months.
Population: All patients were considered to be evaluable for adverse events. Frequency of treatment related adverse events equal to or more than 10% graded to be either 1 (mild), 2 (moderate),3 (severe), 4 (life-threatening).
Measure: Number; unit: participants
Arm/Group | Treatment (Tivozanib)
Number analyzed (Participants) | 58
participants
  Fatigue | 28
  Hypertension | 25
  Nausea | 18
  Diarrhea | 16
  Vomiting | 9
  Hyperglycemia | 12
  Headache | 13
  Lymphopenia | 11
  Anorexia | 12
  Hoarseness | 11
  Aspartate aminotransferase increased | 10
  GGT increased | 10
  Dyspnea | 9
  Cough | 9
  Constipation | 8
  Alkaline phosphatase increase | 9
  Thrombocytopenia | 8
  Myalgia | 9
  Oral Mucositis | 6
  Weight loss | 7
  Hyponatremia | 6

7. Post Hoc Outcome: Number of Patients With 0-3 VEGFR3 Protein Expression and Time in Days on Treatment
Description: Tissue from biopsy will be collected during screening and proteins (VEGFR3) will be evaluated to see if there is a correlation with patient response to treatment.
  VERGFR = vascular endothelial growth factor receptor
  To determine if there was a correlation between response to Tivozanib and VEGFR expression, immunohistochemical (IHC) analysis on archival tumor tissue was performed. We performed standard IHC and applied combined intensity score (from 0 to 3) for antigen expression and proportional score of 0-3 for the cells that were positive. For antigen expression, 0 was no staining, +1 being 1-25% staining, +2 being 26-50% staining and +3 being 50% or greater staining. Number of patients with VEGFR1 expression was correlated with time patients were on treatment in days.
Time Frame: Tissue collected during screening process, prior to first treatment and response measured until 350 days.
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Treatment (Tivozanib)
Number analyzed (Participants) | 40
participants
  VEGFR3 Group 0 : 0 days | 26
  VEGFR3 Group 0 : 50 days | 14
  VEGFR3 Group 0 : 100 days | 7
  VEGFR3 Group 0 : 150 days | 4
  VEGFR3 Group 0 : 200 days | 2
  VEGFR3 Group 0 : 250 days | 2
  VEGFR3 Group 0 : 300 days | 2
  VEGFR3 Group 0 : 350 days | 0
  VEGFR3 Group +1 : 0 days | 7
  VEGFR3 Group +1 : 50 days | 6
  VEGFR3 Group +1 : 100 days | 2
  VEGFR3 Group +1 : 150 days | 1
  VEGFR3 Group +1 : 200 days | 0
  VEGFR3 Group +1 : 250 days | 0
  VEGFR3 Group +1 : 300 days | 0
  VEGFR3 Group +1 : 350 days | 0
  VEGFR3 Group +2 : 0 days | 2
  VEGFR3 Group +2 : 50 days | 1
  VEGFR3 Group +2 : 100 days | 0
  VEGFR3 Group +2 : 150 days | 0
  VEGFR3 Group +2 : 200 days | 0
  VEGFR3 Group +2 : 250 days | 0
  VEGFR3 Group +2 : 300 days | 0
  VEGFR3 Group +2 : 350 days | 0
  VEGFR3 Group +3 : 0 days | 5
  VEGFR3 Group +3 : 50 days | 1
  VEGFR3 Group +3 : 100 days | 1
  VEGFR3 Group +3 : 150 days | 0
  VEGFR3 Group +3 : 200 days | 0
  VEGFR3 Group +3 : 250 days | 0
  VEGFR3 Group +3 : 300 days | 0
  VEGFR3 Group +3 : 350 days | 0

8. Post Hoc Outcome: Number of Patients With 0-3 PDGFR Alpha and PDGFR Beta Protein Expression and Time in Days on Treatment
Description: Tissue from biopsy will be collected during screening and proteins (PDGFR alpha and PDGFR beta) will be evaluated to see if there is a correlation with patient response to treatment.
  PDGFR= Platelet derived growth factor receptor
  To determine if there was a correlation between response to Tivozanib and PDGFR expression, immunohistochemical (IHC) analysis on archival tumor tissue was performed. We performed standard IHC and applied combined intensity score (from 0 to 3) for antigen expression and proportional score of 0-3 for the cells that were positive. For antigen expression, 0 was no staining, +1 being 1-25% staining, +2 being 26-50% staining and +3 being 50% or greater staining. Number of patients with PDGFR alpha and PDGFR beta expression was correlated with time patients were on treatment in days.
Time Frame: Tissue collected during screening process, prior to first treatment and response measured until 350 days.
Population: 3 patients were not evaluable due to withdrawal tivozanib within the first 14 days of treatment. Not all patients treated on study provided tissue or had sufficient tissue to be analyzed for PDGFR expression. No patients showed PDGFR alpha +1 or +3 expression.
Measure: Number; unit: participants
Arm/Group | Treatment (Tivozanib)
Number analyzed (Participants) | 40
participants
  PDGFR alpha Group 0 : 0 days | 38
  PDGFR alpha Group 0 : 50 days | 21
  PDGFR alpha Group 0 : 100 days | 10
  PDGFR alpha Group 0 : 150 days | 5
  PDGFR alpha Group 0 : 200 days | 2
  PDGFR alpha Group 0 : 250 days | 2
  PDGFR alpha Group 0 : 300 days | 2
  PDGFR alpha Group 0 : 350 days | 0
  PDGFR alpha Group+2 : 0 days | 2
  PDGFR alpha Group+2 : 50 days | 1
  PDGFR alpha Group+2 : 100 days | 0
  PDGFR alpha Group+2 : 150 days | 0
  PDGFR alpha Group+2 : 200 days | 0
  PDGFR alpha Group+2 : 250 days | 0
  PDGFR alpha Group+2 : 300 days | 0
  PDGFR alpha Group+2 : 350 days | 0
  PDGFR beta Group 0 : 0 days | 26
  PDGFR beta Group 0 : 50 days | 14
  PDGFR beta Group 0 : 100 days | 7
  PDGFR beta Group 0 : 150 days | 4
  PDGFR beta Group 0 : 200 days | 2
  PDGFR beta Group 0 : 250 days | 2
  PDGFR beta Group 0 : 300 days | 2
  PDGFR beta Group 0 : 350 days | 0
  PDGFR beta Group +1 : 0 days | 7
  PDGFR beta Group +1 : 50 days | 6
  PDGFR beta Group +1 : 100 days | 2
  PDGFR beta Group +1 : 200 days | 1
  PDGFR beta Group +1 : 150 days | 0
  PDGFR beta Group +1 : 250 days | 0
  PDGFR beta Group +1 : 300 days | 0
  PDGFR beta Group +1 : 350 days | 0
  PDGFR beta Group +2 : 0 days | 2
  PDGFR beta Group +2 : 50 days | 1
  PDGFR beta Group +2 : 100 days | 0
  PDGFR beta Group +2 : 150 days | 0
  PDGFR beta Group +2 : 200 days | 0
  PDGFR beta Group +2 : 250 days | 0
  PDGFR beta Group +2 : 300 days | 0
  PDGFR beta Group +2 : 350 days | 0
  PDGFR beta Group +3 : 0 days | 5
  PDGFR beta Group +3 : 50 days | 1
  PDGFR beta Group +3 : 100 days | 1
  PDGFR beta Group +3 : 150 days | 0
  PDGFR beta Group +3 : 200 days | 0
  PDGFR beta Group +3 : 250 days | 0
  PDGFR beta Group +3 : 300 days | 0
  PDGFR beta Group +3 : 350 days | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected over 2 years and 10 months
Arm/Group | Treatment (Tivozanib)
All-Cause Mortality (participants affected / at risk) | 49/58
Serious Adverse Events (participants affected / at risk) | 26/58
Other Adverse Events (participants affected / at risk) | 58/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Tivozanib) (N=58)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 2 (2)
Clinical deterioration (General disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Death NOS (General disorders) | 2 (2)
Localized edema (General disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Pain (General disorders) | 4 (4)
Lung infection (Infections and infestations) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3)
Sepsis (Infections and infestations) | 1 (1)
Ejection fraction decreased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle cramps (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Myelitis (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 3 (3)
Hydronephrosis (Renal and urinary disorders) | 1 (1)
Urinary tract obstuction (Renal and urinary disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumorthorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Tivozanib) (N=58)
Anemia (Blood and lymphatic system disorders) | 19 (26)
Leukocytosis (Blood and lymphatic system disorders) | 5 (5)
Hypothyroidism (Endocrine disorders) | 6 (6)
Hyperthyroidism (Endocrine disorders) | 6 (7)
Blurred vision (Eye disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 9 (10)
Constipation (Gastrointestinal disorders) | 10 (10)
Diarrhea (Gastrointestinal disorders) | 19 (24)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 7 (9)
Nausea (Gastrointestinal disorders) | 21 (25)
Oral pain (Gastrointestinal disorders) | 2 (2)
Stomach pain (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 13 (17)
Edema - limbs (General disorders) | 3 (3)
Fatigue (General disorders) | 29 (38)
Fever (General disorders) | 5 (9)
Gait disturbance (General disorders) | 2 (2)
Non-cardiac chest pain (General disorders) | 2 (2)
Pain (General disorders) | 16 (20)
Urinary tract infection (Infections and infestations) | 5 (5)
Activated partial thromboplastin time prolonged (Investigations) | 20 (24)
Alanine aminotransferase increased (Investigations) | 10 (10)
Alkaline phosphatase increased (Investigations) | 16 (23)
Aspartate aminotransferase increased (Investigations) | 18 (19)
Blood bilirubin increased (Investigations) | 5 (9)
Creatinine increased (Investigations) | 2 (2)
Ejection fraction decreased (Investigations) | 5 (5)
GGT increased (Investigations) | 16 (19)
INR increased (Investigations) | 10 (11)
Lymphocyte count decreased (Investigations) | 28 (34)
Platelet count decreased (Investigations) | 12 (14)
Weight loss (Investigations) | 8 (8)
White blood cell decreased (Investigations) | 4 (4)
Anorexia (Metabolism and nutrition disorders) | 13 (16)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 27 (49)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 31 (46)
Hypocalcemia (Metabolism and nutrition disorders) | 5 (6)
Hypoglycemia (Metabolism and nutrition disorders) | 4 (4)
Hypokalemia (Metabolism and nutrition disorders) | 13 (20)
Hyponatremia (Metabolism and nutrition disorders) | 18 (23)
Hypophosphatemia (Metabolism and nutrition disorders) | 10 (18)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (12)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (13)
Dizziness (Nervous system disorders) | 3 (3)
Headaches (Nervous system disorders) | 15 (15)
Memory impairment (Nervous system disorders) | 2 (2)
Urinary Frequency (Renal and urinary disorders) | 4 (4)
Proteinuria (Renal and urinary disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (14)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 14 (16)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 11 (12)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (4)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2)
Hypertension (Vascular disorders) | 29 (42)
Hypotension (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes